CLINICAL TRIAL: NCT04455685
Title: Prevalence of Self-reported Premenstrual Syndrome and Analysis of Somatic and Psychoemotional Symptoms in Brazilian Women Aged 20 to 49 Years
Brief Title: Prevalence of Self-reported Premenstrual Syndrome and Analysis of Somatic and Psychoemotional Symptoms
Acronym: LB2007
Status: Completed | Type: Observational
Sponsor: Libbs Farmacêutica LTDA (Industry)
Responsible Party: Sponsor
Other Study IDs: LB2007
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: anonymised data collection — The population of the present study corresponds to a sample of previous market research. Data from participants from the five main regions of Brazil (North, Northeast, Midwest, South, Southeast) will be selected at random and according to the sample size calculation.

SUMMARY:
In Brazil there are few published studies that study, the prevalence, symptoms and the population's knowledge about the premenstrual syndrome of women of reproductive age, and that correlate these data with the sociodemographic conditions of these women. In addition, given the complexity of the diagnosis of PMS, the prevalence of PMS in the Brazilian female population may be lower than the self-reported and published in these works, since not all women who believe they suffer from PMS fully comply with the criteria contemplated in the consensus for diagnosis of PMS. In this sense, this study aims to analyze the prevalence and intensity of frequent symptoms of PMS reported by the Brazilian female population. The information generated with this study may help to rethink behaviors to improve the health and quality of life of these women, as well as offer tools for decision making related to the need for early and effective treatment of PMS, whose disorders are associated with both the fall present and future quality of life for women, as well as all of their family, social and professional coexistence.

DETAILED DESCRIPTION:
In Brazil and Latin America there are still few published studies that study, the prevalence, symptoms and the population's knowledge about the premenstrual syndrome of women of reproductive age, and that correlate these data with the sociodemographic, socioeconomic and sociocultural conditions of these women .

In the investigator's view, this study brings value not only to contribute to the understanding and demystification of PMS by society in general, but also for the professionals who assist these women. The data currently used in Brazil, and which are frequently used to guide public health policies, are mostly the result of research carried out in other countries, and which may not correspond to the national reality.

The information generated with this study may help to rethink behaviors to improve the health and quality of life of these women, at this stage in which comprehensive attention to the health and needs of this population should be given, often providing contraceptive methods that offer, as a benefit relief of symptoms related to PMS. The data from this research may also offer tools for decision making related to the need for early and effective treatment of PMS, whose disorders are associated with both the decrease in the present and future quality of life for the woman, as well as all of her family life, social and professional.

ELIGIBILITY:
Inclusion Criteria:

* Data from questionnaires that integrate the anonymous secondary database generated in the period between 20/02/2019 and 03/20/2020, of female participants aged between 20 and 49 years, in which all necessary information has been filled out according to the participant's profile.

Exclusion Criteria:

* The present study does not include exclusion criteria

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the present study corresponds to a sample of previous market research. Data from participants from the five main regions of Brazil (North, Northeast, Midwest, South, Southeast) will be selected at random and according to the sample size calculation.
Sampling Method: Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
sociodemographic data | 4 months
  Data from at least 1022 (one thousand and twenty-two) women, aged between 20 and 49 years old, living in the five regions of Brazil will be retrieved at random. This information will be organized in a data collection form developed for this study.
somatic and psychoemotional premenstrual symptoms data | 4 months
  data related to somatic and psychoemotional premenstrual symptoms, with their intensity measured by a 4-point Likert scale (0 = none; 1 = mild; 2 = moderate; 3 = severe), degree of interference of these symptoms in daily life and whether the participants would take contraceptives as a method of treating PMS. These data will be organized in a data collection form prepared for this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusto Theodoro de Figueiredo, São Paulo, Brazil